CLINICAL TRIAL: NCT03119597
Title: A Randomized, Double-blind, Placebo-controlled Study Investigating the Effects of Blueberry Anthocyanin on Cognitive Functioning and Mood in Adolescents.
Brief Title: An Investigation Into the Effects of Blueberry Anthocyanin on Cognitive Functioning and Mood in Adolescents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Wild Blueberry Association of North America (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor in Behavioral Neuroscience, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RDG002
Record Dates: First submitted 2017-03-23; First posted 2017-04-18 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Depression
Keywords: low mood, depression
MeSH Terms: conditions — Depression; Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: participants will be assigned to either a Placebo or Blueberry (treatment) drink, in parallel for the duration of the study
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the researchers will be aware of which participants are receiving treatment or placebo. Participants and their parents will be debriefed on the last test day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Formulation containing approximately 4.79g Fructose+ 4.52g Glucose+ 45mg Vitamin C
  Interventions: Dietary Supplement: Placebo
- Wild Blueberry Power-13g (Experimental): Formulation containing approximately 250mg of anthocyanin+ 4.79g Fructose+ 4.52g Glucose+ 45mg Vitamin C
  Interventions: Dietary Supplement: Wild Blueberry Powder-13g

INTERVENTIONS:
Dietary Supplement: Wild Blueberry Powder-13g — Formulation containing approximately 250mg of anthocyanin+ 4.79g Fructose+ 4.52g Glucose+ 45mg Vitamin C
  Arms: Wild Blueberry Power-13g
Dietary Supplement: Placebo — Formulation containing approximately 4.79g Fructose+ 4.52g Glucose+ 45mg Vitamin C
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a 4-week dietary intervention with wild blueberry powder can have an effect on cognitive performance in participants aged between 13-17.

DETAILED DESCRIPTION:
Interventions: Flavonoid drink and a matched placebo will be used in this study. Flavonoid drink will contain approximately, 13g of freeze dried wild blueberry powder, containing 250mg of anthocyanin flavonoid, mixed with 170ml water and flavored with 30ml 'Rock's Organic Orange Squash' as it has a low flavonoid content. The placebo drink will contain placebo powder matched for vitamin C (45mg), glucose (4.52g) and fructose (4.79g), mixed with 170ml of water and 30ml 'Rock's Organic Orange Squash'. Participants will be randomly allocated to either placebo or treatment. Participants will be instructed to consume the drink every morning for 4 weeks. The powder will be prepared and sealed in opaque packets. Participants will be provided with 2 weeks worth of supplies at baseline and then in week 2. Parents will be provided with instructions on how to prepare the drinks in addition to supplies such as opaque straws and containers. Assessment of left-over product will be conducted in 2 weeks to allow for continued compliance verification.

Procedure: the study comprises of a screen and four visits, including a familiarization week and 2 test visits.

1. Screening: Once a school has indicated interest in aiding with this trial, participants will be given a brief overview of the study and asked to complete a set of questionnaires regarding their mood and general health to confirm suitability for participating in this study. The questionnaires include Mood and Feeling Questionnaire (MFQ) and Revised Child Anxiety and Depression Scale (RCADS).Participants who score 27 or above (depressed) and score 14 or below (healthy) on the MFQ will be invited to participate in the second part of the study. Parents of the participants meeting the criteria will then be contacted to ascertain that each interested volunteer and parents are willing to participate for the entire duration of the study and to schedule their familiarization visit.
2. Familiarization Visit: Volunteers and parents will be invited to volunteers' first visit at the location of volunteers' choice (Nutritional Psychology Unit at the University of Reading or volunteers' school) where participants will receive a detailed explanation of the study by the participating research associate and will be asked to sign the informed consent form before any study procedure starts. A log will be kept identifying all participants having signed the informed consent form (ICF) and the participant will be allocated a participant number. Once consent has been given, the participants will then be asked to complete the EPIC Food Frequency Questionnaire so that background flavonoid intakes can be measured prior to the start of the intervention, Rumination Response Scale (RRS) and a General health questionnaire. Participants intelligence quotient (IQ) will be assessed using The Wechsler Abbreviated Scale of Intelligence (WASIII). Parents will also be asked to complete questionnaires, regarding children mood and behaviors, including the Parent version of MFQ, RCADS and attention deficit hyperactivity disorder (ADHD) Rating Scale-IV. Finally, participants will be given training on the cognitive test battery (tasks outlined below) that will be used during the study to reduce the chances of 'practice' adversely affecting performance on subsequent test days.
3. Test Visits (Weeks 0, 2 and 4): All of these sessions will be held at times that suit participants' individual needs. The timings of the testing sessions will be consistent for each participant over the 4 weeks. Upon arrival, participants will be asked of any adverse events and any issues with compliance. Participants will then complete the battery of cognitive tasks consisting of (i) Modified Eriksen Flanker task, (ii) The Keep track task (KTT) and (iii)The Controlled Oral Word Association Test (COWAT), in addition to completing the daily mood measure Positive and Negative Affect Schedule (PANAS). Additionally, the last test session (week 4) participants and parents' will once again be asked to complete the MFQ, RCADS and RRS mentioned above.

Participants may stop the study treatment without stating any reason at any time during the study. In addition, a participant will be withdrawn from the study if a volunteer or parents request a discontinuation, participant exhibits a serious adverse event to any component of the test product, an illness emerges and/or the investigator's opinion is that withdrawal is appropriate and in the best interest of the participant. If a participant withdraws from the study, participants will be encouraged to make a final visit as soon as possible, irrespective of the reason for withdrawal, to complete a final battery of cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy volunteers as proven by medical history and/or physical examination and of all ethnicity and socioeconomic status
* Participants at risk of depression or healthy as assessed by MFQ (score 27 or above and score 14 or below)
* Able to get a parent or guardian to give signed written informed consent in addition to they themselves giving informed assent

Exclusion Criteria:

* Use of complementary and alternative medicine
* History of metabolic disorder, diabetes, or other medical conditions.
* Participants using medications that might affect the outcome measures, such as antidepressant and sleeping medication.
* Participants who score between 14 and 27 on the MFQ.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Change in Working Memory performance | 0, 2 and 4 weeks
  Keep tract task: measuring working memory performance
Change in Mood | 0, 2 and 4 weeks
  measured by use of PANAS
Change in verbal fluency | 0, 2 and 4 weeks
  Controlled oral word association task: measuring working memory performance
Change in Cognitive Accuracy | 0, 2 and 4 weeks
  Modified Flanker Task: measuring accuracy
Change in reaction time | 0, 2 and 4 weeks
  Modified Flanker Task: measuring reaction time
Change in Depression | 0 and 4 weeks
  measured by use of MFQ
Change in Anxiety | 0 and 4 weeks
  measured by use of RCADS

SECONDARY OUTCOMES:
Change in Rumination | 0 and 4 week
  Measured using Rumination Response Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes